CLINICAL TRIAL: NCT03737929
Title: Comparison of the Efficacy of Hybrid Ablative Therapy for Patients with Persistent Atrial Fibrillation Versus Conventional Catheter Ablation
Brief Title: Hybrid Therapy and Heart Team for Atrial Fibrillation
Acronym: HT2AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0449
Record Dates: First submitted 2018-10-31; First posted 2018-11-13 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: Epicardial surgical ablation; Percutaneous endocardial catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid ablation procedure (Experimental): In the hybrid ablation procedure, the epicardial surgical ablation procedure will be combined with percutaneous endocardial catheter ablation procedure in a single step procedure.
  Interventions: Procedure: Hybrid ablation
- Percutaneous endocardial catheter ablation procedure (Active Comparator): In the percutaneous catheter ablation arm, the procedure will be performed according to the current guidelines (pulmonary vein isolation, linear ablation and fragmented potentials ablation if needed, with the achievement of sinus rhythm during the procedure being the optimal endpoint).
  Interventions: Procedure: Percutaneous catheter ablation

INTERVENTIONS:
Procedure: Hybrid ablation — In the hybrid ablation arm, the epicardial surgical ablation procedure will be combined with percutaneous endocardial catheter ablation procedure in a single step procedure (same operative time). During the endocardial approach, the isolation of the pulmonary veins and the posterior box will be checked and completed if necessary. Then additional ablation will be performed for atrial tachycardia or ongoing persisting atrial fibrillation (AF) according the same lesions setup or stepwise protocol than the conventional arm
  Arms: Hybrid ablation procedure
Procedure: Percutaneous catheter ablation — In the percutaneous catheter ablation arm, the procedure will be performed according to the current guidelines (pulmonary vein isolation, linear ablation and fragmented potentials ablation if needed, with the achievement of sinus rhythm during the procedure being the optimal endpoint. Any atrial tachycardia will be mapped and ablated as well (DC shock performed otherwise).
  Arms: Percutaneous endocardial catheter ablation procedure

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia with a prevalence ranging from 5% over 60 years old to 17% after 85 years old. Besides hemodynamical compromises and occurrence of heart failure, stroke remains the most feared complication related to AF with a risk increased by 5-fold.

Catheter ablation with the aim of pulmonary veins isolation (PVI) has evolved as a standardized treatment option in paroxysmal AF (PAF), supported by the current guidelines. However, due to advanced electrical and structural remodeling, catheter ablation for persistent AF is rather disappointing with a limited success rate, at least after a single procedure. Due to these shortcomings, minimally invasive thoracoscopic surgical techniques have gained attention with good results in persistent AF patients. Comparison between thoracoscopic surgical ablation and catheter ablation have shown that surgical ablation was associated with higher success rates, less redo procedures but also with higher complication rates. The main issue with surgical ablation is the difficulty to check the ablation lines and pulmonary vein isolation, which are the cornerstones for achieving good long-term results.

Hybrid therapy, combining both epicardial surgical and endocardial catheter ablation is expected to be the most effective technique. It would avoid incomplete lesions or incomplete pulmonary vein isolation, and would provide complete lesion set. Hybrid therapy of AF has been compared with mini-invasive surgical ablation of AF, showing a significant higher rate of sinus rhythm achievement in the hybrid therapy group. However, no comparative clinical trials data are currently available in the setting of persistent AF comparing hybrid ablation and conventional catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

* To have a history of symptomatic persistent atrial fibrillation (AF) (continuous AF lasting 7 days or more) or long-standing persistent AF (continuous AF lasting for more than 12 months)
* To be refractory to or intolerant to at least one class I (flecainide / propafenone) or III (sotalol / amiodarone) antiarrhythmic drug,
* To be at least 18 years of age,
* To agree to participate (signature of the informed consent)

Exclusion Criteria:

* A previous AF ablation procedure,
* A longstanding persistent AF > 3 years,
* A paroxysmal AF
* AF consecutive to electrolyte imbalance, thyroid disease, or other reversible non-cardiovascular cause,
* Presence of left atrial appendage (LAA) thrombus,
* Left atrial size ≥ 70ml/m² on transthoracic echocardiogram (TTE),
* Left ventricular ejection fraction < 35%,
* Cardiac surgery (other than AF treatment) planned within 12 months,
* Contra-indication to heparin and/or oral anticoagulation
* Contra-indication to transoesophageal echocardiogram (TEE)
* Carotid stenosis > 80%,
* Active infection or sepsis
* Pleural adhesions,
* Elevated hemi diaphragm
* Proven and untreated sleep apnoea syndrome,
* Occurrence of a cerebrovascular accident (CVA) or a transient ischemic attack (TIA) during the past 6 months,
* History of blood clotting abnormalities
* Indication for a permanent dual antiplatelet therapy
* History of thoracic radiation,
* History of myocarditis or pericarditisHistory of cardiac tamponade,
* History of thoracotomy or cardiac surgery,
* Body-mass-index > 40 kg/m2,
* Significant lung dysfunction
* Contra-indication to anesthesia
* Patient with chronic obstructive pulmonary disease (COPD)
* Pregnancy,
* Life expectancy less than 12 months,
* Adults protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation (AF)/Atrial tachycardia (AT) recurrence | 12 months
  occurrence of at least one episode of AF/AT > 30 seconds in any ECG or Holter tracing (absence or presence)

SECONDARY OUTCOMES:
AF/AT recurrence or major complication | 12 months
  Percentage of patients developing a recurrence of AF/AT or a major complication (related to the procedure or related to AF/AT)
Major complication related to the procedure | 12 months
  Percentage of patients developing a major complication related to the procedure
Major complication related to AF/AT | 12 months
  Percentage of patients developing a major complication related to AF/AT
Any complication (major or minor) | 12 months
  Percentage of patients developing any complication (major or minor) related to the procedure or related to AF/AT
Redo-procedure | 12 months
  Percentage of patients requiring a redo-procedure (new ablation in left atrium)
Cardioversion | 12 months
  Percentage of patients requiring a cardioversion
Number of hospitalizations | 12 months
  Number of hospitalizations for AF/AT recurrence or complications related to AF/AT or to the procedure
Duration of the hospitalization | 1 month
  Mean duration of the hospitalization for AF ablation
Radiation exposure time | 12 months
  Radiation exposure time (expressed in minutes) per patient. In case of redo-ablation during the follow-up, the total exposure time of the two first and the redo procedure will be totalized.
Radiation exposure dosage | 12 months
  Radiation exposure dosage per patient. In case of redo-ablation during the follow-up, the total exposure dosage of the two first and the redo procedure will be totalized.
Antiarrhythmic drugs | 12 months
  Percentage of patients requiring class I (flecainide ou propafenone) or III (sotalol ou amiodarone) antiarrhythmic drugs
Electrophysiological success | Day 0
  Percentage of patients considered as reaching electrophysiological success, i.e. isolation of pulmonary veins and posterior box after epicardial surgical ablation. The validation will be performed during catheter ablation: isolation will be validated if there an entrance block in the posterior wall and in the pulmonary veins.
Evolution of quality of life | Between baseline to 12 months
  Evolution of quality of life using the Canadian Cardiovascular Society Severity in Atrial Fibrillation (CCS-SAF) scale. Symptom severity, physical and emotional components of quality of life, general well-being, and health care consumption related to AF are evaluated by this scale. The scale ranges from 0 to 4, corresponding to 0=no effect on functional quality of life to 4=a severe effect on life quality.
ICER | 12 months
  The incremental cost-effectiveness ratio (ICER) of hybrid ablation versus catheter ablation, including long term evaluation with MARKOV modelling
ICUR | 12 months
  The incremental Cost-Utility Ratio (ICUR) of hybrid ablation versus catheter ablation, including long term evaluation with MARKOV modelling
Production costs | during the surgical procedure
  Production costs of the two strategies using the micro-costing approach

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Maury, MD, Principal Investigator — University Hospital of Toulouse
Locations (3):
- France (3):
  - Cardiology-rytmology, Paris
  - CHU Toulouse, Hôpital Rangueil, Toulouse
  - Cardiology-rytmology service, Toulouse

IPD SHARING:
Plan to Share IPD: No